CLINICAL TRIAL: NCT00333177
Title: Developmental Processes in Schizophrenic Disorders: Cognitive Remediation, Medication Adherence, and Work Outcome in Recent-Onset Schizophrenia
Brief Title: Psychosocial Therapy and Risperidone Treatment in Work Performance in Recent-Onset Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Keith Nuechterlein, Ph.D., Prinicipal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH037705-06 (NIH); R01MH037705 (NIH); DAHBR AD-P (Registry Identifier: WHO ICTRP)
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Schizophrenia
Keywords: Schizoaffective Disorder, Depressed Type; Schizophreniform Disorder; First-Episode Schizophrenia; Supported Employment; Cognitive Remediation; Health Behavior Training; Antipsychotic Medication
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cog Remediation, risperidone injection (Experimental): Participants will receive cognitive remediation training plus risperidone, administered via injection.
  Interventions: Behavioral: Cognitive remediation training (CT); Drug: Risperidone, administered via injection (RLAI)
- Healthy Behavior Training, risperidone injection (Active Comparator): Participants will receive health behavior training plus risperidone, administered via injection.
  Interventions: Behavioral: Healthy behavior training (HBT); Drug: Risperidone, administered via injection (RLAI)
- Cog Remediation, oral risperidone (Experimental): Participants will receive cognitive remediation training plus risperidone administered orally.
  Interventions: Behavioral: Cognitive remediation training (CT); Drug: Risperidone, administered orally (Oral Ris)
- Healthy Behavior Training, oral risperidone (Active Comparator): Participants will receive health behavior training plus risperidone administered orally.
  Interventions: Behavioral: Healthy behavior training (HBT); Drug: Risperidone, administered orally (Oral Ris)

INTERVENTIONS:
Behavioral: Cognitive remediation training (CT) — Cognitive remediation training includes computerized cognitive training plus learning skills group.
  Arms: Cog Remediation, oral risperidone; Cog Remediation, risperidone injection
Behavioral: Healthy behavior training (HBT) — Healthy behavior training includes group skills training in nutrition, exercise, and relaxation.
  Arms: Healthy Behavior Training, oral risperidone; Healthy Behavior Training, risperidone injection
Drug: Risperidone, administered orally (Oral Ris) — Oral risperidone at dosage judged optimal by treating psychiatrist
  Other Names: Risperdal
  Arms: Cog Remediation, oral risperidone; Healthy Behavior Training, oral risperidone
Drug: Risperidone, administered via injection (RLAI) — Risperidone in injectable form every 2 weeks, starting with 25 mg and adjusted as needed
  Other Names: Risperdal Consta
  Arms: Cog Remediation, risperidone injection; Healthy Behavior Training, risperidone injection

SUMMARY:
This study will determine the effectiveness of various combinations of psychosocial therapy and risperidone treatment in improving work or school performance in people with first-episode schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a chronic, severe, and disabling brain disorder. People with schizophrenia often experience hallucinations, delusions, thought disorders, and movement disorders. These symptoms make it difficult to maintain a job, participate in school, and keep up self-care. Proper treatment of first-episode schizophrenia may increase the chances of controlling disease progression on a long-term basis. Antipsychotic medications, such as risperidone, and psychosocial treatments, such as cognitive enhancement training and health behavior training, are common, effective treatments for schizophrenia. This study will determine the effectiveness of various combinations of psychosocial therapy and risperidone treatment in improving work or school performance in people with first-episode schizophrenia.

Participants in this open label study will be randomly assigned to receive one of the following four combinations of an antipsychotic medication and a psychosocial treatment: cognitive enhancement training plus oral risperidone; cognitive enhancement training plus long-acting injectable risperidone; health behavior training plus oral risperidone; or health behavior training plus long-acting injectable risperidone. Cognitive enhancement training will entail 2 hours per week of computer-assisted training targeted at improving attention, memory, and problem-solving skills. Additionally, participants will attend a weekly 1-hour group meeting to learn how to apply these skills to work and school situations. Health behavior training will involve 3 hours per week of relaxation training, nutrition education, and physical exercise to enhance wellness. Participants assigned to receive oral risperidone will receive their medication in pill form at the dosage determined to be optimal by the study psychiatrist. Participants assigned to receive injectable risperidone will be given one injection every 2 weeks. Dosages will start at 25 mg per injection and will be adjusted as needed.

Treatment will continue for 1 year following dosage stabilization, which typically occurs 2 to 3 months following study entry. For the first 6 months, participants assigned to receive health behavior training will attend study visits once a week and participants assigned to receive cognitive enhancement training will attend study visits once a week. For the final 6 months, all participants will attend study visits twice weekly. At each visit, participants will receive their assigned psychosocial treatment; attend group therapy; meet with a case manager for counseling and assessment of symptoms, work functioning, and social functioning; and meet with a psychiatrist to monitor medication response. Additional cognitive and health behavior measures will be taken every 6 months to assess treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, schizoaffective disorder (depressed type), or schizophreniform disorder
* First major episode of psychotic symptoms occurred within 2 years prior to study entry

Exclusion Criteria:

* Neurological disorder or injury (e.g., encephalitis, epilepsy, traumatic brain injury)
* Mental retardation (e.g., premorbid intelligence quotient (IQ) less than 70)
* Significant alcohol or substance use during last 6 months
* Unable to complete research measures in English
* Any condition that may make risperidone use medically inadvisable

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2006-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith H. Nuechterlein, PhD, Principal Investigator — University of California, Los Angeles, Department of Psychiatry and Biobehavioral Sciences
Locations (1):
- Semel Institute for Neuroscience and Human Behavior at UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nuechterlein KH, Ventura J, Subotnik KL, Gretchen-Doorly D, Turner LR, Casaus LR, Luo J, Boucher ML, Hayata JN, Bell MD, Medalia A. A randomized controlled trial of cognitive remediation and long-acting injectable risperidone after a first episode of schizophrenia: improving cognition and work/school functioning. Psychol Med. 2022 Jun;52(8):1517-1526. doi: 10.1017/S0033291720003335. Epub 2020 Sep 28. PMID 32981534
- [Derived] Subotnik KL, Casaus LR, Ventura J, Luo JS, Hellemann GS, Gretchen-Doorly D, Marder S, Nuechterlein KH. Long-Acting Injectable Risperidone for Relapse Prevention and Control of Breakthrough Symptoms After a Recent First Episode of Schizophrenia. A Randomized Clinical Trial. JAMA Psychiatry. 2015 Aug;72(8):822-9. doi: 10.1001/jamapsychiatry.2015.0270. PMID 26107752

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 32 patients who were enrolled in the study dropped out during the initial medication stabilization period prior to the start of randomized treatment resulting in 60 being assigned to the randomized treatments.
Groups:
- CT - RLAI: Participants will receive cognitive remediation training (CT) plus injectable, long-acting risperidone (RLAI).
  Cognitive remediation: Cognitive remediation training includes computerized cognitive training plus learning skills group.
  Risperidone, administered via injection: Risperidone in injectable form every 2 weeks, starting with 25 mg and adjusted as needed
  Individual Placement and Support: Supported education/employment
- HBT - RLAI: Participants will receive health behavior training (HBT) plus injectable, long-acting risperidone (RLAI).
  Health behavior training: Health behavior training includes group skills training in nutrition, exercise, and relaxation.
  Risperidone, administered via injection: Risperidone in injectable form every 2 weeks, starting with 25 mg and adjusted as needed
  Individual Placement and Support: Supported education/employment
- CT - Oral Ris: Participants will receive cognitive remediation training (CT) plus risperidone administered orally (Oral Ris).
  Cognitive remediation: Cognitive remediation training includes computerized cognitive training plus learning skills group.
  Risperidone, administered orally: Oral risperidone at dosage judged optimal by treating psychiatrist
  Individual Placement and Support: Supported education/employment
- HBT - Oral Ris: Participants will receive health behavior training (HBT) plus risperidone administered orally (Oral Ris).
  Health behavior training: Health behavior training includes group skills training in nutrition, exercise, and relaxation.
  Risperidone, administered orally: Oral risperidone at dosage judged optimal by treating psychiatrist
  Individual Placement and Support: Supported education/employment
Period: Overall Study
Arm/Group | CT - RLAI | HBT - RLAI | CT - Oral Ris | HBT - Oral Ris
Started | 12 | 17 | 17 | 14
Received Intervention | 12 | 16 | 16 | 12
Completed | 12 | 16 | 16 | 12
Not Completed | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- CT - RLAI: Participants will receive cognitive remediation training plus injectable, long-acting risperidone.
  Cognitive remediation: Cognitive remediation training includes computerized cognitive training plus learning skills group.
  Risperidone, administered via injection: Risperidone in injectable form every 2 weeks, starting with 25 mg and adjusted as needed
  Individual Placement and Support: Supported education/employment
- HBT - RLAI: Participants will receive health behavior training plus injectable, long-acting risperidone.
  Health behavior training: Health behavior training includes group skills training in nutrition, exercise, and relaxation.
  Risperidone, administered via injection: Risperidone in injectable form every 2 weeks, starting with 25 mg and adjusted as needed
  Individual Placement and Support: Supported education/employment
- CT - Oral Ris: Participants will receive cognitive remediation training plus risperidone administered orally.
  Cognitive remediation: Cognitive remediation training includes computerized cognitive training plus learning skills group.
  Risperidone, administered orally: Oral risperidone at dosage judged optimal by treating psychiatrist
  Individual Placement and Support: Supported education/employment
- HBT - Oral Ris: Participants will receive health behavior training plus risperidone administered orally.
  Health behavior training: Health behavior training includes group skills training in nutrition, exercise, and relaxation.
  Risperidone, administered orally: Oral risperidone at dosage judged optimal by treating psychiatrist
  Individual Placement and Support: Supported education/employment
- Total: Total of all reporting groups
Arm/Group | CT - RLAI | HBT - RLAI | CT - Oral Ris | HBT - Oral Ris | Total
Number analyzed (Participants) | 12 | 17 | 17 | 14 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.7 (2.9) | 22.1 (4.6) | 21.3 (3.1) | 20.8 (3.3) | 21.9 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5 | 4 | 14
  Male | 10 | 14 | 12 | 10 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 9 | 6 | 25
  Not Hispanic or Latino | 8 | 11 | 8 | 8 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 3 | 2 | 1 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 7 | 5 | 2 | 17
  White | 6 | 8 | 10 | 10 | 34
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 17 | 17 | 14 | 60

OUTCOME MEASURES:

1. Primary Outcome: Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: Values presented here are the changes in MCCB Overall Composite T scores from baseline to 12 months, with higher values representing better outcome. Raw test scores are used to generate T-scores and then the seven MCCB domains are combined to generate an Overall Composite T score. MCCB Overall Composite T scores have a mean in the general population of 50 with a standard deviation of 10. Thus, a positive change of 5 T scores is an improvement of half a standard deviation.
Time Frame: Measured at baseline and 12 months
Population: All participants with MCCB outcome data.
Measure: Mean (Standard Error); unit: T scores
Arm/Group | CT - RLAI | HBT - RLAI | CT - Oral Ris | HBT - Oral Ris
Number analyzed (Participants) | 12 | 16 | 16 | 12
T scores | 6.7 (1.9) | 0.9 (1.6) | 3.9 (1.6) | 5.9 (1.9)
Statistical Analysis 1: Comparison: CT - RLAI vs HBT - RLAI vs CT - Oral Ris vs HBT - Oral Ris; A priori hypothesis was that CT would be superior to HBT and that RLAI would enhance this effect; Test type: Superiority; p < 0.03, ANCOVA — P value is for CT-HBT X RLAI-Oral Ris interaction; Covaried baseline value of dependent variable

2. Primary Outcome: Work/School Functioning (Global Functioning Scale: Role)
Description: Change in role functioning from baseline to the 6 month point (rated on a scale from 1= Extreme Role Dysfunction to 10 = Superior Role Functioning) is presented here.
Time Frame: Baseline to 6 months
Population: Participants who received services from the supported education/employment specialist
Measure: Mean (Standard Deviation); unit: Changes on a 10-point scale
Arm/Group | CT - RLAI | HBT - RLAI | CT - Oral Ris | HBT - Oral Ris
Number analyzed (Participants) | 10 | 12 | 15 | 11
Changes on a 10-point scale | 2.90 (2.56) | 0.92 (2.75) | 1.27 (2.76) | -0.82 (2.93)
Statistical Analysis 1: Comparison: CT - RLAI vs HBT - RLAI vs CT - Oral Ris vs HBT - Oral Ris; 2 X 2 ANOVA was calculated. A priori hypotheses were that LAI would be superior to oral risperidone and that CT would be superior to health behavior training (HBT) based on main effects; Test type: Superiority; p < .02, ANCOVA — P-value is for each main effect. A priori threshold for statistical significance was p<0.05 for each main effect; Baseline value of dependent variable was covaried

3. Primary Outcome: Average Medication Non-adherence
Description: 5-point scale (1 = best adherence, 5= nonadherent) based on pill counts, Medication Event Monitoring System (MEMS) cap readings, plasma assays, and psychiatrist judgements for oral risperidone and timing of injections for long-acting injectable risperidone. Averaged over medication study participation.
Time Frame: Averaged over study participation (up to 12 months)
Population: A priori hypothesis was that long-acting injectable risperidone would result in better medication adherence than oral risperidone, so CT and HBT groups were merged within each medication administration condition.
Measure: Mean (Standard Deviation); unit: units on a 5-point scale
Groups:
- RLAI: Participants will receive risperidone, administered via injection: Risperidone in injectable form every 2 weeks, starting with 25 mg and adjusted as needed
  For this study aim, only the medication comparison is involved, so the cognitive training and Health Behaviors Training groups are combined within this medication condition. Participants will receive either cognitive remediation or healthy behaviors training plus risperidone administered by injection. All participants received individual Placement and Support: Supported education/employment
- Oral Ris: Risperidone, administered orally: Oral risperidone at dosage judged optimal by treating psychiatrist.
  For this study aim, only the medication comparison is involved, so the cognitive training and Health Behaviors Training groups are combined within this medication condition. Participants will receive either cognitive remediation or healthy behaviors training plus risperidone administered orally.All participants received individual Placement and Support: Supported education/employment
Arm/Group | RLAI | Oral Ris
Number analyzed (Participants) | 28 | 27
units on a 5-point scale | 1.0 (0.1) | 1.9 (0.7)
Statistical Analysis 1: Comparison: RLAI vs Oral Ris; A priori hypothesis was that RLAI would lead to less medication non-adherence than Oral Ris; Test type: Superiority; p = .001, t-test, 2 sided; Mean Difference (Final Values) = .84, 95% CI 2-sided [.57 to 1.10]

4. Primary Outcome: Work/School Functioning (Global Functioning Scale: Role)
Description: Changes in role functioning from baseline to 12 months. Ratings on a 10-point scale with 10 being best.
Time Frame: Baseline to 12 months
Population: Participants who received services from the Individual Placement and Support specialist.
Measure: Mean (Standard Deviation); unit: Changes on a 10-point scale
Arm/Group | CT - RLAI | HBT - RLAI | CT - Oral Ris | HBT - Oral Ris
Number analyzed (Participants) | 10 | 13 | 14 | 11
Changes on a 10-point scale | 2.70 (2.67) | 1.69 (2.66) | 2.43 (2.44) | 0.18 (3.19)
Statistical Analysis 1: Comparison: CT - RLAI vs HBT - RLAI vs CT - Oral Ris vs HBT - Oral Ris; 2 X 2 ANOVA was calculated. A priori hypotheses were that CT would be superior to HBT and that RLAI would be superior to Oral Ris; Test type: Superiority; p < .05, ANCOVA — P-value is for CT vs. HBT main effect; Baseline value of dependent variable was covaried

5. Secondary Outcome: Work Behavior Inventory (WBI) Quality of Work/School Performance
Description: Change in rating on quality of work/school performance based on patient, employer, and/or teacher reports. The Quality of Work rating at baseline was subtracted from the same rating at 12 mos. Higher scores are better outcome.
Time Frame: Baseline to 1 year
Population: This measure could be rated only for individuals who were in school or working at baseline and at 12 months, so it proved not to be useful due to the infrequent return to school or work by baseline.
Measure: Mean (Standard Deviation); unit: score on a rating scale
Arm/Group | CT - RLAI | HBT - RLAI | CT - Oral Ris | HBT - Oral Ris
Number analyzed (Participants) | 2 | 6 | 8 | 2
score on a rating scale | -6.5 (31.8) | 8.8 (34.0) | -3.4 (17.4) | 0.0 (33.9)
Statistical Analysis 1: Comparison: CT - RLAI vs HBT - RLAI vs CT - Oral Ris vs HBT - Oral Ris; Test type: Superiority; p = 0.55, ANOVA

6. Secondary Outcome: Maintenance of Work/School Attendance
Description: Modified Work Section of the Social Adjustment Scale (SAS) was used to calculate the total number of weeks in school or competitive work. Range of possible values is 0 to 52, with higher numbers being better outcome.
Time Frame: 12 months
Population: Participants who were served by the Individual Placement and Support specialist
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | CT - RLAI | HBT - RLAI | CT - Oral Ris | HBT - Oral Ris
Number analyzed (Participants) | 12 | 16 | 16 | 12
weeks | 35.4 (21.2) | 24.4 (19.8) | 26.7 (20.0) | 12.0 (12.8)
Statistical Analysis 1: Comparison: CT - RLAI vs HBT - RLAI vs CT - Oral Ris vs HBT - Oral Ris; Test type: Superiority; p < 0.02, ANOVA — A priori hypotheses were that CT would be superior to HBT and that RLAI would be superior to Oral Ris; 2 X 2 ANOVA was computed

7. Secondary Outcome: Exacerbation or Relapse of Psychotic Symptoms
Description: Dichotomous measure: Presence of any of 3 psychotic relapse or exacerbation categories scored from the Brief Psychiatric Rating Scale (BPRS) occurring after randomization and until end of study participation (up to 12 months post baseline). BPRS was administered every two weeks throughout study participation.
Time Frame: Occurence after randomization and until end of study participation (up to 12 mos.)
Population: A priori hypothesis was that RLAI would lead to fewer psychotic exacerbations/relapses than Oral Ris. No effect of CT vs. HBT was hypothesized, so CT and HBT conditions were merged within each medication administration condition.
Measure: Number; unit: participants
Arm/Group | RLAI | Oral Ris
Number analyzed (Participants) | 28 | 28
participants | 2 | 10
Statistical Analysis 1: Comparison: RLAI vs Oral Ris; Chi-square of frequencies of relapse vs. non-relapse were calculated, with a priori hypothesis that RLAI would be superior to Oral Ris; Test type: Superiority; p < 0.01, Chi-squared; df = 1

8. Secondary Outcome: Retention in Treatment
Description: Days after randomization that a participant continued to receive at least the assigned CT or HBT psychosocial treatment. If a participant needed to end the assigned medication condition (RLAI vs. Oral Ris), they continued in the psychosocial treatment so this outcome focused on the days in the assigned psychosocial treatment. Possible range is 1 to 365, with higher being a better outcome.
Time Frame: 12 months
Population: All participants who received Individual Placement and Support
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CT - RLAI | HBT - RLAI | CT - Oral Ris | HBT - Oral Ris
Number analyzed (Participants) | 12 | 16 | 16 | 12
days | 359.7 (8.1) | 352.2 (26.9) | 332.4 (38.8) | 348.3 (28.4)
Statistical Analysis 1: Comparison: CT - RLAI vs HBT - RLAI vs CT - Oral Ris vs HBT - Oral Ris; Test type: Superiority; p < .05, ANOVA — 2 X 2 ANOVA calculated. P-value is for main effect of RLAI vs. Oral Ris

9. Secondary Outcome: Awareness of Illness, as Assessed by the Scale to Assess Unawareness of Mental Disorder, Revised Version (SUMD-R)
Description: Rating scale based on clinician's interview of patient to determine level of lack of awareness of having a mental disorder. Range is from 1 (Aware) to 5 (Unaware), so lower scores indicate better outcome.
Time Frame: 12 months after randomization
Population: All participants with SUMD-R data at 12-month point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CT - RLAI | HBT - RLAI | CT - Oral Ris | HBT - Oral Ris
Number analyzed (Participants) | 4 | 7 | 6 | 4
score on a scale | 1.25 (0.50) | 3.29 (1.80) | 2.00 (1.67) | 3.75 (0.96)
Statistical Analysis 1: Comparison: CT - RLAI vs HBT - RLAI vs CT - Oral Ris vs HBT - Oral Ris; Test type: Superiority; p < .02, ANOVA — 2 X 2 ANOVA computed. P-value is for main effect of CT vs. HBT

10. Secondary Outcome: Change in Motivation for Work/School
Description: The Work Motivation scale is a factor score from the Work Personality Profile. The Work Personality Profile is a set of ratings based on interviewing the participant. Scores at each occasion can range from 8 to 32, with higher indicating better motivation. Scores reported here are changes from baseline to 12 months, which could range from -24 to 24 with higher being better.
Time Frame: Baseline to 12 months
Population: Participants in school or jobs at baseline and 12 months, which allows change in Work Personality Profile ratings to be assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CT - RLAI | HBT - RLAI | CT - Oral Ris | HBT - Oral Ris
Number analyzed (Participants) | 7 | 6 | 9 | 5
score on a scale | 3.7 (2.3) | 1.2 (4.6) | -2.4 (7.4) | -1.9 (6.5)
Statistical Analysis 1: Comparison: CT - RLAI vs HBT - RLAI vs CT - Oral Ris vs HBT - Oral Ris; Test type: Superiority; p = .053, ANOVA — 2 X 2 ANOVA computed. P-value is for RLAI vs. Oral Ris main effect

11. Secondary Outcome: Change in Coping Strategies
Description: Coping Response Inventory, which rates extent to which active coping strategies were used after a significant stressful life event. Range of possible scores is 1 to 4. Higher scores are better.
Time Frame: Baseline to 12 months
Population: Participants with Coping Response Inventories completed for a comparable stressful life event at baseline and 12 months. This was so rare in practice that this outcome was not feasible to evaluate.
Arm/Group | CT - RLAI | HBT - RLAI | CT - Oral Ris | HBT - Oral Ris
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | CT - RLAI | HBT - RLAI | CT - Oral Ris | HBT - Oral Ris
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/16 | 3/16 | 1/12
Other Adverse Events (participants affected / at risk) | 5/12 | 5/16 | 11/16 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT - RLAI (N=12) | HBT - RLAI (N=16) | CT - Oral Ris (N=16) | HBT - Oral Ris (N=12)
psychiatric hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) — psychiatric hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT - RLAI (N=12) | HBT - RLAI (N=16) | CT - Oral Ris (N=16) | HBT - Oral Ris (N=12)
BMI increase normal/overweight to Obese (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 5 (5) | 0 (0) — Increase in BMI from normal/overweight to any Obese category
LDL or Triglyceride increase (Cardiac disorders) | 1 (1) | 1 (1) | 4 (4) | 5 (5) — increase from normal to high in either LDL or Triglyceride
TD early signs (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Early signs of mild tardive dyskinesia
Prolactin related symptom (Endocrine disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2) — Symptom related to prolactin level

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No